CLINICAL TRIAL: NCT06937853
Title: The Effect of Genetic Polymorphisms on the Response to Preoperative Non-Steroidal Anti-Inflammatory Drugs in the Management of Endodontic Postoperative Pain
Brief Title: Effect of Genetic Polymorphisms on Response to Preoperative NSAIDs in Endodontic Postoperative Pain Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ertuğrul karataş, Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/297
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain
Keywords: Endodontics Genetic Polymorphism NSAIDs Preoperative Analgesia Pain Sensitivity
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Diclofenac

STUDY DESIGN:
Intervention Model Description: This study adopts a parallel assignment model in which participants are randomly allocated into three groups: diclofenac sodium, ibuprofen, or placebo. Each participant receives a single dose of the assigned medication prior to root canal treatment. The primary aim is to evaluate the effectiveness of preoperative NSAIDs in reducing postoperative endodontic pain.
  Additionally, the study explores whether genetic variations in drug-metabolizing enzymes affect individual responses to these medications. By analyzing these genetic differences, the study aims to determine their potential influence on postoperative pain levels, ultimately contributing to more personalized pain management approaches in dental practice.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ibuprofen Group (Experimental): Participants in this arm will receive a single oral dose of 600 mg ibuprofen prior to the endodontic procedure. This intervention is intended to evaluate the preemptive analgesic effect of ibuprofen in the control of postoperative endodontic pain.
  Interventions: Drug: Ibuprofen 600 mg
- diclofenac sodium (Experimental): Participants in this arm will receive a single oral dose of 100 mg diclofenac sodium prior to the endodontic procedure. This intervention is intended to assess the preemptive analgesic efficacy of diclofenac sodium in controlling postoperative endodontic pain.
  Interventions: Drug: diclofenac sodium
- placebo (Placebo Comparator): Participants in this arm will receive a single oral dose of a placebo tablet, identical in appearance to the active drugs, prior to the endodontic procedure. This group serves as a control to assess the true analgesic efficacy of the active interventions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen 600 mg — A single oral dose of 600 mg ibuprofen will be administered prior to the endodontic procedure to evaluate its preemptive analgesic effect on postoperative dental pain.
  Arms: Ibuprofen Group
Drug: diclofenac sodium — A single oral dose of 100 mg diclofenac sodium will be administered to participants in the Diclofenac Sodium Group prior to the endodontic procedure. This intervention is designed to assess the preemptive analgesic efficacy of diclofenac sodium in the control of postoperative dental pain.
  Arms: diclofenac sodium
Drug: Placebo — A single oral dose of a placebo tablet, identical in appearance to the active drugs, will be administered to participants in the Placebo Group prior to the endodontic procedure. This group serves as the control to evaluate the true analgesic efficacy of the active interventions.
  Arms: placebo

SUMMARY:
This study aims to evaluate the influence of genetic polymorphisms on the effectiveness of preoperative non-steroidal anti-inflammatory drugs (NSAIDs) in managing postoperative pain following endodontic treatment. Participants will receive standard preoperative NSAIDs before undergoing root canal therapy, and their pain responses will be assessed. Genetic analysis will be performed to investigate possible associations between drug response and individual gene variations. The study seeks to improve personalized approaches in endodontic pain management.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18 and 65 years
2. Vital mandibular molar teeth diagnosed with symptomatic apical periodontitis
3. ASA physical status classification I or II
4. Preoperative VAS pain score greater than 50
5. No known genetic disorders (e.g., Down syndrome, congenital insensitivity to pain)

Exclusion Criteria:

1. Patients classified as ASA III or higher
2. Pregnant women or those suspected of being pregnant
3. Presence of root canal curvature greater than 25° (Schilder classification)
4. Patients with generalized periodontitis
5. Presence of periodontal pockets deeper than 3 mm in the affected tooth
6. History of systemic disease or known allergies
7. Patients with diagnosed psychiatric or psychological disorders
8. Presence of swelling, sinus tract, or preoperative tenderness on palpation
9. Patients with bruxism
10. Presence of resorption in the affected tooth
11. Use of analgesic or anti-inflammatory drugs within 12 hours prior to the procedure
12. Teeth with root fractures, ankylosis, or pathological mobility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-08-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | 7 days after treatment
  Pain intensity will be evaluated using the Visual Analog Scale (VAS). The scale ranges from 0 mm (no pain) to 100 mm (worst imaginable pain). A higher score indicates a worse outcome (more severe pain).
  Patients will be asked to mark their pain level at 6 hours, 12 hours, 24 hours, and on postoperative days 2 (48 hours), 3 (72 hours), 5, and 7 following endodontic treatment.
  The mean VAS scores at each time point will be analyzed and compared between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ertugrul Karatas, Prof. Dr., Principal Investigator — Ataturk University, Faculty of Dentistry, Department of Endodontics
Locations (1):
- Ataturk University, Faculty of Dentistry, Department of Endodontics, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] AlRahabi MK. Predictors, prevention, and management of postoperative pain associated with nonsurgical root canal treatment: A systematic review. J Taibah Univ Med Sci. 2017 May 9;12(5):376-384. doi: 10.1016/j.jtumed.2017.03.004. eCollection 2017 Oct. PMID 31435267